CLINICAL TRIAL: NCT01898741
Title: Cone-beam CT Guided Stereotactic Radiation Therapy for Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, M. van Vulpen, Professor, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCU-12-628
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Radiotherapy; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irradiation (Experimental): 24 Gy in 3 fractions
  Interventions: Radiation: 24 Gy in 3 fractions

INTERVENTIONS:
Radiation: 24 Gy in 3 fractions

SUMMARY:
Pancreatic cancer has a very poor survival, due to late diagnosis and lack of sufficient treatment options for locally advanced tumors and metastasized patients. High dose radiotherapy with small margins seems feasible with current technical possibilities, e.g. by fiducial guided stereotactic radiotherapy. In this study, we want to evaluate safety and technical feasibility for cone beam CT guided stereotactic radiotherapy for locally advanced pancreatic carcinoma.

DETAILED DESCRIPTION:
Objective of the study:

To determine safety and technical feasibility of stereotactic radiotherapy for locally advanced pancreatic carcinoma

Study design:

Pilot study to determine safety and feasibility

Study population:

Patients with locally advanced pancreatic carcinoma, without distant metastasis

Intervention:

Patients will undergo endoscopic fiducial marker placement, and patients will get a custom-made individual corset. Radiotherapy will be delivered in three fractions of 8 Gy on an outpatient basis.

Primary study outcome:

The main study endpoint will be safety of the procedure, expressed in proportion of patients experiencing treatment-induced toxicity grade 3 or more according to the CTC-AE 4.0 due to the complete procedure within 90 days of the last radiation.

Secondary study outcome:

Other study parameters will be technical feasibility, treatment response, quality of life, overall survival, progression free survival, and rate of possible secondary resections

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Increased severe toxicity may occur due to the intervention, but treatment related toxicity should be limited due to strict dose constraints to the organs at risk (e.g. duodenum, stomach). Potential benefits may be pain relief, due to local control of the tumor, and a prolonged survival.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced pancreatic tumors (stage III) or medically inoperable patients with pancreatic cancer (stage I, II, or III)
* Not eligible for operation with curative intent
* >18 years
* Written informed consent

Exclusion Criteria:

* WHO performance status 3-4
* Expected life span <3 months
* Previous chemotherapy, pancreatic surgery or pancreatic radiotherapy
* Exclusion criteria for contrast enhanced MRI and/or CT scan, following the protocol of the department of radiology UMCU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Safety | 90 days of last irradiation
  Safety of the procedure, expressed in proportion of patients experiencing treatment-induced toxicity grade 3 or more according to the CTC-AE 4.0 due to the complete procedure within 90 days of the last radiation

CONTACTS AND LOCATIONS:
Overall Officials: M. van Vulpen, Prof MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Heerkens HD, van Vulpen M, Erickson B, Reerink O, Intven MP, van den Berg CA, Molenaar IQ, Vleggaar FP, Meijer GJ. MRI guided stereotactic radiotherapy for locally advanced pancreatic cancer. Br J Radiol. 2018 Nov;91(1091):20170563. doi: 10.1259/bjr.20170563. Epub 2018 Jul 31. PMID 30063383